CLINICAL TRIAL: NCT03024099
Title: Effects of Weekly Hippotherapy Frequency on Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Alessandra Vidal Prieto, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 50019415.3.0000.0030
Record Dates: First submitted 2017-01-08; First posted 2017-01-18 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2017-01

CONDITIONS: Cerebral Palsy
Keywords: hippotherapy Gross Motor Function Functional performance.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hippotherapy once a week (Experimental): Hippotherapy once a week;
  Interventions: Other: Hippotherapy once a week
- Hippotherapy twice a week (Experimental): hippotherapy twice a week
  Interventions: Other: Hippotherapy twice a week

INTERVENTIONS:
Other: Hippotherapy once a week — Hippotherapy once a week
  Arms: Hippotherapy once a week
Other: Hippotherapy twice a week — Hippotherapy twice a week
  Arms: Hippotherapy twice a week

SUMMARY:
The hippotherapy is considered a therapeutic modality that provides numerous benefits in the rehabilitation process and has often been recommended by doctors for children with cerebral palsy. Despite being in frank ascent, this therapy still lacks scientific evidence. Objectives: To analyze and compare the effects of hippotherapy program, often 1 or 2 days a week in gross motor function, trunk balance and functional performance of children with cerebral palsy.

DETAILED DESCRIPTION:
Study characterized by a controlled experiment with a sample of 24 children, aged between 2 and 4 years, were randomly divided into control group (CG), with 9 participants, with the use of 1 to week and experimental group, also with 11 participants, 2 times a week intervention. The call followed protocol and took place once or twice a week lasting 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 to 6 years of age with diagnosis of Cerebral Palsy, besides medical, physiotherapeutic and psychological referral with indication of the practice of Hippotherapy
* Children classified with GMFCS levels 2, 3, 4 or 5
* Understanding, agreement and signing of the Free and Informed Consent Form
* Understanding, agreement and signing of the Free and Informed Assent Term, when applicable
* Possibility to participate in a riding program 1 or 2 times a week for a period of 16 weeks
* Conduct traditional physiotherapy concomitantly 1 or 2 times a week

Exclusion Criteria:

* Presence of associated syndromes or structural deformities that make Hippotherapy impossible
* Present seizures without medication control
* Does not have enough hip joint amplitude for riding (about 20 degrees of abduction)
* To have an invasive or surgical procedure during the study
* Have previously participated in an Equine Therapy program

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Effects of weekly frequency of hippotherapy on gross motor function through GMFM (gross motor function measurement) of children with cerebral palsy. | one year
  GMFM - quantitative scale assessing 5 dimensions of motor development.
Effects of weekly frequency of hippotherapy on functional performance through the Pediatric Disability Inventory (PEDI) of children with cerebral palsy. | one year
  PEDI Inventory - quantitative scale that evaluates the functional performance, among others, for self care, mobility and social function.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alemdaroglu E, Yanikoglu I, Oken O, Ucan H, Ersoz M, Koseoglu BF, Kapicioglu MI. Horseback riding therapy in addition to conventional rehabilitation program decreases spasticity in children with cerebral palsy: A small sample study. Complement Ther Clin Pract. 2016 May;23:26-9. doi: 10.1016/j.ctcp.2016.02.002. Epub 2016 Feb 13. PMID 27157954
- [Background] Borgi M, Loliva D, Cerino S, Chiarotti F, Venerosi A, Bramini M, Nonnis E, Marcelli M, Vinti C, De Santis C, Bisacco F, Fagerlie M, Frascarelli M, Cirulli F. Effectiveness of a Standardized Equine-Assisted Therapy Program for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Jan;46(1):1-9. doi: 10.1007/s10803-015-2530-6. PMID 26210515
- [Background] Jang B, Song J, Kim J, Kim S, Lee J, Shin HY, Kwon JY, Kim YH, Joung YS. Equine-Assisted Activities and Therapy for Treating Children with Attention-Deficit/Hyperactivity Disorder. J Altern Complement Med. 2015 Sep;21(9):546-53. doi: 10.1089/acm.2015.0067. Epub 2015 Jul 13. PMID 26167851
- [Background] Park J, Lee S, Lee D. The effects of horseback riding simulator exercises on the muscle activity of the lower extremities according to changes in arm posture. J Phys Ther Sci. 2015 Sep;27(9):2731-2. doi: 10.1589/jpts.27.2731. Epub 2015 Sep 30. PMID 26504280
- [Background] Lee DK, Kim EK. The influence of horseback riding training on the physical function and psychological problems of stroke patients. J Phys Ther Sci. 2015 Sep;27(9):2739-41. doi: 10.1589/jpts.27.2739. Epub 2015 Sep 30. PMID 26504283
- [Background] Angsupaisal M, Visser B, Alkema A, Meinsma-van der Tuin M, Maathuis CG, Reinders-Messelink H, Hadders-Algra M. Therapist-Designed Adaptive Riding in Children With Cerebral Palsy: Results of a Feasibility Study. Phys Ther. 2015 Aug;95(8):1151-62. doi: 10.2522/ptj.20140146. Epub 2015 Apr 23. PMID 25908525
- [Background] Kang KY. Effects of mechanical horseback riding on the balance ability of the elderly. J Phys Ther Sci. 2015 Aug;27(8):2499-500. doi: 10.1589/jpts.27.2499. Epub 2015 Aug 21. PMID 26355558
- [Background] Cho SH, Kim JW, Kim SR, Cho BJ. Effects of horseback riding exercise therapy on hormone levels in elderly persons. J Phys Ther Sci. 2015 Jul;27(7):2271-3. doi: 10.1589/jpts.27.2271. Epub 2015 Jul 22. PMID 26311966
- [Background] Kim SR, Cho SH, Kim JW, Lee HC, Brienen M, Cho BJ. Effects of horseback riding exercise therapy on background electroencephalograms of elderly people. J Phys Ther Sci. 2015 Jul;27(7):2373-6. doi: 10.1589/jpts.27.2373. Epub 2015 Jul 22. PMID 26311985
- [Background] Lee N, Park S, Kim J. Effects of hippotherapy on brain function, BDNF level, and physical fitness in children with ADHD. J Exerc Nutrition Biochem. 2015 Jun;19(2):115-21. doi: 10.5717/jenb.2015.15061209. Epub 2015 Jun 30. PMID 26244130
- [Background] Flores FM, Dagnese F, Mota CB, Copetti F. Parameters of the center of pressure displacement on the saddle during hippotherapy on different surfaces. Braz J Phys Ther. 2015 May-Jun;19(3):211-7. doi: 10.1590/bjpt-rbf.2014.0090. Epub 2015 Jun 12. PMID 26083600
- [Background] Earles JL, Vernon LL, Yetz JP. Equine-assisted therapy for anxiety and posttraumatic stress symptoms. J Trauma Stress. 2015 Apr;28(2):149-52. doi: 10.1002/jts.21990. Epub 2015 Mar 17. PMID 25782709
- [Background] Lee CW, Kim SG, An BW. The effects of horseback riding on body mass index and gait in obese women. J Phys Ther Sci. 2015 Apr;27(4):1169-71. doi: 10.1589/jpts.27.1169. Epub 2015 Apr 30. PMID 25995581
- [Background] Kwon JY, Chang HJ, Yi SH, Lee JY, Shin HY, Kim YH. Effect of hippotherapy on gross motor function in children with cerebral palsy: a randomized controlled trial. J Altern Complement Med. 2015 Jan;21(1):15-21. doi: 10.1089/acm.2014.0021. Epub 2014 Dec 31. PMID 25551626
- [Background] Temcharoensuk P, Lekskulchai R, Akamanon C, Ritruechai P, Sutcharitpongsa S. Effect of horseback riding versus a dynamic and static horse riding simulator on sitting ability of children with cerebral palsy: a randomized controlled trial. J Phys Ther Sci. 2015 Jan;27(1):273-7. doi: 10.1589/jpts.27.273. Epub 2015 Jan 9. PMID 25642090
- [Background] Park ES, Rha DW, Shin JS, Kim S, Jung S. Effects of hippotherapy on gross motor function and functional performance of children with cerebral palsy. Yonsei Med J. 2014 Nov;55(6):1736-42. doi: 10.3349/ymj.2014.55.6.1736. PMID 25323914
- [Background] Kwon JY, Chang HJ, Lee JY, Ha Y, Lee PK, Kim YH. Effects of hippotherapy on gait parameters in children with bilateral spastic cerebral palsy. Arch Phys Med Rehabil. 2011 May;92(5):774-9. doi: 10.1016/j.apmr.2010.11.031. PMID 21530725
- [Background] McGibbon NH, Benda W, Duncan BR, Silkwood-Sherer D. Immediate and long-term effects of hippotherapy on symmetry of adductor muscle activity and functional ability in children with spastic cerebral palsy. Arch Phys Med Rehabil. 2009 Jun;90(6):966-74. doi: 10.1016/j.apmr.2009.01.011. PMID 19480872
- [Background] Tseng SH, Chen HC, Tam KW. Systematic review and meta-analysis of the effect of equine assisted activities and therapies on gross motor outcome in children with cerebral palsy. Disabil Rehabil. 2013 Jan;35(2):89-99. doi: 10.3109/09638288.2012.687033. Epub 2012 May 26. PMID 22630812